CLINICAL TRIAL: NCT00539773
Title: Phase II Trial of Concurrent Administration of Intravesical BCG & Interferon in the Treatment and Prevention of Recurrence of Superficial Transitional Carcinoma of the Urinary Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2011-073
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Transitional Carcinoma of Urinary Bladder
MeSH Terms: interventions — Interferons

INTERVENTIONS:
Drug: BCG, Interferon — Chemotherapy

SUMMARY:
Phase II Trial of concurrent administration of intravesical BCG & Interferon in the treatment and prevention of recurrence of superficial transitional carcinoma of the urinary bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with superficial transitional carcinoma of the urinary bladder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Efficacy | overall

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia